CLINICAL TRIAL: NCT04297969
Title: Detection of Hyperopia by Photoscreener GoCheckKids With Glow Fixation Device
Brief Title: Hyperopia Detection GCK With Glow Fixation
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ABCD GCK Glow
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-03

CONDITIONS: Amblyopia Bilateral; Hyperopia of Both Eyes; Astigmatism Bilateral; Accommodation Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- GCK Glow fixation: Patients screened with GoCheck Kids flash concentrated iPhone 7+
  Interventions: Diagnostic Test: objective pediatric vision screen "GCK glow fixation"

INTERVENTIONS:
Diagnostic Test: objective pediatric vision screen "GCK glow fixation" — 2-axis, smart phone flash concentrated photoscreen using novel, low-detail, color glow fixation device
  Other Names: objective pediatric vision screening GCK glow fixation

SUMMARY:
"GoCheck Kids" has added to its iPhone 7+ smart phone with flash concentrator a non-accommodating glow box fixation target. In pediatric eye patients, the "GCK" with glow box is compared to cycloplegic refraction as well as School Bus Accommodation-relaxing skiascopy, "2WIN" photoscreener and "Retinomax."

DETAILED DESCRIPTION:
Patients undergoing comprehensive pediatric eye exam were screened with "GoCheck Kids" iPhone 7+ flash concentrated photoscreener with new, non-accommodating glow fixation target are well as "Adaptica 2WIN" photoscreener and "Retinomax" auto refraction all without drops before cycloplegia examination.

Reason for examination, visual acuity, ocular alignment and degree of amblyopia were specifically noted.

Refractive amblyopia risk factors utilizing "AAPOS 2003" and "AAPOS 2013" uniform guidelines were used to validate each screening method.

Patients for whom cycloplegia exam yielded at least 0.5 diopters hyperopia were compared to determine the ability of each screening tool to detect hyperopia.

ELIGIBILITY:
Inclusion Criteria:

* Patients having comprehensive pediatric eye examination

Exclusion Criteria:

* Patients with only one eye

Ages: 1 Month to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with a range of refractive errors including high hyperopia and astigmatism in a pediatric ophthalmology referral practice.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
2003 and 2013 AAPOS Uniform Amblyopia Risk Factor (ARF) prevalence | 1 week
  presence of refractive risk factors (anisometropia >1.50D, hyperopia > 3.5D, Astigmatism >1.50D, myopia more than 3D

SECONDARY OUTCOMES:
Amblyopia | 1 week
  Presence of amblyopia defined by decreased visual acuity with normal anatomy plus amblyopia risk factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Alaska Children's EYE & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data via website
Supporting Information: CSR
Time Frame: 1 month from now
Access Criteria: Study website
URL: http://www.abcd-vision.org/references/index.html

REFERENCES:
- [Background] Racano E, Alessi S, Pertile R. Comparison of 2Win and plusoptiX A12R refractometers with Retinomax handheld autorefractor keratometer. J AAPOS. 2019 Oct;23(5):276.e1-276.e5. doi: 10.1016/j.jaapos.2019.05.017. Epub 2019 Sep 17. PMID 31539614
- [Background] Arnold SL, Arnold AW, Sprano JH, Arnold RW. Performance of the 2WIN Photoscreener With "CR" Strabismus Estimation in High-Risk Patients. Am J Ophthalmol. 2019 Nov;207:195-203. doi: 10.1016/j.ajo.2019.04.016. Epub 2019 May 9. PMID 31077668
- [Background] Peterseim MMW, Rhodes RS, Patel RN, Wilson ME, Edmondson LE, Logan SA, Cheeseman EW, Shortridge E, Trivedi RH. Effectiveness of the GoCheck Kids Vision Screener in Detecting Amblyopia Risk Factors. Am J Ophthalmol. 2018 Mar;187:87-91. doi: 10.1016/j.ajo.2017.12.020. Epub 2018 Jan 2. PMID 29305313
- [Background] Arnold RW, O'Neil JW, Cooper KL, Silbert DI, Donahue SP. Evaluation of a smartphone photoscreening app to detect refractive amblyopia risk factors in children aged 1-6 years. Clin Ophthalmol. 2018 Aug 23;12:1533-1537. doi: 10.2147/OPTH.S171935. eCollection 2018. PMID 30197499
- [Background] Arnold RW, Arnold AW, Hunt-Smith TT, Grendahl RL, Winkle RK. The Positive Predictive Value of Smartphone Photoscreening in Pediatric Practices. J Pediatr Ophthalmol Strabismus. 2018 Nov 19;55(6):393-396. doi: 10.3928/01913913-20180710-01. Epub 2018 Aug 29. PMID 30160295
- [Background] Levitt AH, Martin SJ, Arnold RW. Performance of Glow Fixation GoCheck Kids and 2WIN Photoscreeners and Retinomax to Uncover Hyperopia. Clin Ophthalmol. 2020 Aug 10;14:2237-2244. doi: 10.2147/OPTH.S256991. eCollection 2020. PMID 32982148
- [Derived] Arnold RW, Beveridge JS, Martin SJ, Beveridge NR, Metzger EJ, Smith KA. Grading Sphero-Cylinder Spectacle Similarity. Clin Optom (Auckl). 2021 Jan 20;13:23-32. doi: 10.2147/OPTO.S289770. eCollection 2021. PMID 33505178